CLINICAL TRIAL: NCT01962974
Title: A Golimumab Phase 3b, Multicenter, Assessment of Intravenous Efficacy in Rheumatoid Arthritis Subjects Who Have Diminished Disease Control Despite Treatment With Infliximab (REMICADE®)
Acronym: REGAIN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Cancelled due to low enrollment
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR102117; CNTO148ART3003 (Other: Janssen Biotech, Inc.); 2013-001809-91 (EudraCT Number)
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Golimumab 2 mg/kg IV (Experimental): Study drug (golimumab 2 mg/kg IV) will be administered as an intravenous (IV) infusion at Weeks 0, 4, 12, 20 and 28.
  Interventions: Biological: Golimumab 2 mg/kg IV

INTERVENTIONS:
Biological: Golimumab 2 mg/kg IV — Study drug (golimumab 2 mg/kg IV) will be administered as an intravenous (IV) infusion at Weeks 0, 4, 12, 20 and 28.

SUMMARY:
This is a Phase 3b, multicenter study of the efficacy of golimumab 2 mg/kg IV in subjects with active rheumatoid arthritis who are receiving methotrexate and have inadequate disease control (defined as an erythrocyte sedimentation rate [ESR]-based Disease Activity Score in 28 joints [DAS28] ≥ 3.2 and ≥ 4 swollen and ≥ 4 tender joints) despite current anti-TNFα therapy with infliximab 2 - 4 mg/kg every 4 weeks, 2 - 5 mg/kg every 5 weeks, 3 - 6 mg/kg every 6 weeks, 3 - 7mg/kg every 7 weeks, or 4 - 8 mg/kg every 8 weeks.

To be eligible for participation, subjects must have previously demonstrated initial and/or temporary improvement in disease signs and symptoms, who have since exhibited a diminished response despite continued treatment. It is estimated that 200 subjects will be enrolled in the study at approximately 85 global sites.

DETAILED DESCRIPTION:
The study employs an open-label "active switch" design that moves subjects from infliximab to golimumab 2 mg/kg IV. In general, subjects eligible for the study include men or women who are currently receiving infliximab in actual clinical practice who are at least 18 years of age with active rheumatoid arthritis, and have previously demonstrated initial and/or temporary improvement in disease signs and symptoms, but now exhibit a diminished response and inadequate disease control despite continued treatment. Subjects must have received infliximab in combination with methotrexate for a minimum of 9 months prior to the first screening visit.

The screening visit will occur sometime between Week -12 and Week -10. Consenting subjects who meet screening criteria will receive their final dose of infliximab at Week -8 as part of actual clinical practice. Golimumab IV treatment, which will be supplied by the sponsor, will be received at Weeks 0, 4, 12, 20, and 28. The primary endpoint is at Week 24, the final efficacy assessment is at Week 32, and a follow-up safety assessment by telephone is at Week 44. There will be a maximum of 36 weeks between the last infliximab infusion at Week -8 and the last infusion of golimumab at Week 28. The duration of study participation is expected to be a maximum of 56 weeks (including the Screening Period, 32 weeks of golimumab treatment and assessment, and a 12-week safety follow-up).

ELIGIBILITY:
Major Inclusion Criteria include (but not limited to):

* Have a diagnosis of Rheumatoid Arthritis (according to the revised 1987 criteria of the American Rheumatism Association).
* Treatment with infliximab and methotrexate for >= 9 months, (with stable doses of methotrexate over last 16 weeks of 7.5 mg/week to 25 mg/week) and (anti-TNFα therapy with infliximab 2 - 4 mg/kg every 4 weeks, 2 - 5 mg/kg every 5 weeks, 3 - 6 mg/kg every 6 weeks, 3 - 7mg/kg every 7 weeks, or 4 - 8 mg/kg every 8 weeks).
* Disease Activity Score 28 (DAS28) ≥ 3.2 based on Erythrocyte Sedimentation Rate (ESR) at Week -8 and Week 0.
* Swollen joint count (SJC) ≥ 4 and tender joint count (TJC) ≥ 4 at Week - 8 and at Week 0.
* Prior response confirmed by physician.

Major Exclusion Criteria include (but not limited to):

* Have a history of latent or active granulomatous infection, including histoplasmosis, or Have a history of latent or active granulomatous infection, including histoplasmosis, or coccidioidomycosis, prior to the first screening visit or during the Screening Period.
* Have had a Bacille Calmette-Guérin (BCG) vaccination within 12 months of screening.
* Have a chest radiograph within 3 months prior to the first administration of study agent that shows an abnormality suggestive of a malignancy or current active infection, including tuberculosis (TB), histoplasmosis, or coccidioidomycosis.
* Have previously received more than 1 of the currently approved subcutaneous (SC) administered anti-TNFα agents, etanercept, certolizumab pegol, golimumab, or adalimumab.
* Are pregnant, nursing, or planning a pregnancy or fathering a child within 6 months after receiving the last administration of the study agent.
* Weight less than 35 kg or greater than 110 kg (less than 77 pounds or greater than 242 pounds).

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (47):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Peoria, Arizona
  - Phoenix, Arizona
  - Fort Smith, Arkansas
  - Fremont, California
  - Fullerton, California
  - Long Beach, California
  - Santa Maria, California
  - Thousand Oaks, California
  - Whittier, California
  - Bridgeport, Connecticut
  - Clearwater, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Coeur d'Alene, Idaho
  - Indianapolis, Indiana
  - South Bend, Indiana
  - Eagan, Minnesota
  - Edina, Minnesota
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Orchard Park, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Wilmington, North Carolina
  - Dayton, Ohio
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Myrtle Beach, South Carolina
  - Hixson, Tennessee
  - Jakson, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Arlington, Virginia
  - Spokane, Washington
  - Glendale, Wisconsin
- Canada (5):
  - Victoria, British Columbia
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - Montreal, Quebec
  - Rimouski

REFERENCES:
- See also: A Golimumab Phase 3b, Multicenter, Assessment of Intravenous Efficacy in Rheumatoid Arthritis Subjects Who Have Diminished Disease Control Despite Treatment with Infliximab (REMICADE ®) REGAIN — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=4785&filename=CR102117_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated early due to low recruitment; only 7 participants were enrolled.
Groups:
- Golimumab: Participants received golimumab 2 milligram per kilogram (mg/kg) intravenously (IV) at Weeks 0, 4, 12, 20, and 28.
Period: Overall Study
Arm/Group | Golimumab
Started | 7
Completed | 0
Not Completed | 7
Not completed — Study termination | 7

BASELINE CHARACTERISTICS:
Arm/Group | Golimumab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 20 (ACR20) Response at Week 24
Description: The ACR 20 Response is defined as greater than or equal to (>=) 20 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and erythrocyte sedimentation rate (ESR).
Time Frame: Week 24
Population: Due to early study termination, data for this outcome measure was not collected and therefore the analyses could not be conducted.
Arm/Group | Golimumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Participants Who Achieved an ACR 20 Response at Week 24 With Confirmed Presence of Antibodies to Infliximab
Description: The ACR 20 Response is defined as >= 20 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: patient's assessment of pain using VAS (010 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and ESR.
Time Frame: Week 24
Population: as for outcome 1
Arm/Group | Golimumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants Who Acheived ACR 20 Response at Week 24 With Trough Infliximab Levels Below the Lower Limit of Quantification (LLOQ)
Description: as for outcome 2
Time Frame: Week 24
Population: as for outcome 1
Arm/Group | Golimumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Golimumab
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
The primary limitation for this study was the very low enrolment, ie, 7 participants which led to the early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.